CLINICAL TRIAL: NCT03373318
Title: Influence of Albumin on the Development of Acute Renal Dysfunction Associated With Cardiac Surgery Under Extracorporeal Circulation
Brief Title: Influence of Albumin on Acute Renal Dysfunction Associated With Cardiac Surgery Under Extracorporeal Circulation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IIBSP-ALB-2017-72
Record Dates: First submitted 2017-12-11; First posted 2017-12-14 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Serum Albumin, Human; Plasmalyte A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Human Albumin
  Interventions: Drug: Human albumin
- Control (Active Comparator): Plasmalyte
  Interventions: Drug: Plasmalyte

INTERVENTIONS:
Drug: Human albumin — Single dose as a primer for the CEC, in sufficient quantity to reach a concentration of 4% of the total volume of priming.
  Arms: Experimental
Drug: Plasmalyte — The dose and the speed of administration depend on the age, weight, clinical and biological status of the patient and the concomitant treatment. The recommended dose for adults, the elderly and adolescents: from 500 ml to 3 liters / 24 hours.
  Arms: Control

SUMMARY:
Acute renal dysfunction associated with cardiac surgery (DRA-ACC) in our hospital population affects 39% of patients, being an important cause of morbidity and mortality, increasing the need for dialysis and assuming a prolongation of stay in the unit of intensive care, as well as an increase in the economic cost.

In this sense, extracorporeal circulation (CPB) is a clear aggression for renal function due to multiple effects, not entirely known.

Human albumin is sometimes used as part of the priming of the CEC circuit in variable concentration according to published centers and studies, demonstrating benefits on the maintenance of plasma oncotic pressure during the period of ECC, as well as other effects that can protect renal function during this period of renal injury.

Despite the use of albumin in the ECC priming both in Spain and in other countries, there are currently no published studies demonstrating the effect of albumin on renal function administered during CPB in cardiac surgery during the postoperative period. with a high incidence of kidney injury, although there are current studies that confirm a decrease in the incidence of kidney injury in patients with hypoalbuminemia and who undergo heart surgery without extracorporeal circulation.

The hypothesis of this study is based on the potential protective effect of albumin on renal function in patients undergoing heart surgery under CPB, in which there is a high incidence of postoperative hypoalbuminemia.

This study aims to obtain information about the effect that albumin can have in this population of patients with a high incidence of acute renal dysfunction, and if this benefit exists, whether it is significant or not to justify its systematic use.

DETAILED DESCRIPTION:
This study is aimed to analyze the effect of the use of human albumin during ECC on the incidence of ARD-ACC in patients undergoing cardiac surgery with CPB diagnosed according to the KDIGO scale during the first 7 days after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years) scheduled for cardiopulmonary bypass surgery with Glomerular Filtration Rate (GFR) greater than or equal to 60 and left ventricular ejection fraction greater than or equal to 40%

Exclusion Criteria:

* Patients who do not meet the inclusion criteria and those who have a history of allergic reactions to human albumin, as well as those who have received iodinated contrast during the 7 days prior to surgery and pregnant women, will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of DRA-ACC | 7 days
  The incidence of DRA-ACC will be defined according to the KDIGO scale, for which the levels of plasma creatinine (mmol / L) will be determined. The KDIGO scale classify the injury or acute renal failure as stage I, II or III using as reference the creatinine levels.

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Miralles, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided